CLINICAL TRIAL: NCT06475911
Title: Impact of Peri-Operative Hyponatremia on Postoperative Outcomes in Major HPB Surgeries for Cancers
Status: Recruiting | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Cancer-01
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-04

CONDITIONS: Carcinoma
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perioperative Hyponatremia: Perioperative Hyponatremia <135 mEq/L
- No Perioperative Hyponatremia: No Perioperative Hyponatremia, i.e s.sodium >135 mEq/L

SUMMARY:
The present study is being designed to study the impact and predictive nature of perioperative hyponatremia on post operative outcomes in patients undergoing Major HPB surgeries for cancers. Major hepatobiliary-pancreatic surgeries will be defined as follows-

* Pancreaticoduodenectomy,
* Hemihepatectomy or greater with or without caudate lobectomy
* Extrahepatic bile duct resection
* Extended cholecystectomy
* Distal Pancreatectomy with or without splenectomy The primary Objective of the study would be to compare post operative major morbidities and early mortality (<90 day) in major HPB surgeries done for cancer patients with and without peri-operative hyponatremia. (<135mmoL/L). Development of systemic complications and long term outcomes (overall survival and disease free survival) will also be evaluated.

It will be an observational study consisting of both, a retrospective arm and a prospective arm. All consecutive patients undergoing major HPB surgery from 2010 till 30th June 2024 will be included in the study.

DETAILED DESCRIPTION:
Primary objective: To compare post operative major morbidities and early mortality (<90 day) in major HPB surgeries done for cancer in patients with and without peri-operative hyponatremia. (<135mmoL/L)

Secondary objectives: To compare the following in patients undergoing major HPB surgeries for cancer in patients with and without peri-operative hyponatremia (<135mmoL/L)

* Post operative Systemic complications and
* Long term outcomes

  * OS- POD1 till death/ last follow up (30th Sep 2024).
  * DFS- Surgical resection till first detected recurrence of cancer or last follow up (30th Sep 2024) without recurrence.
* Study design- Observational study- Retrospective and prospective.
* Study period- Data collection will be done from time of ethical clearance till 30th June 2024.
* Intervention - None
* Monitoring and assessment- Clinical profile of the patient and symptoms will be serially followed during the patients post operative OPD visits.
* STATISTICAL ANALYSIS:

  1. Continuous variables- with Student t test and Mann Whitney U test as appropriate.
  2. Categorical data - Chi square or Fischer exact test. Besides the above, appropriate analysis will be done at the time of final data analysis.
  3. Significance will be seen at 5 % level (p<0.05).
  4. Adequate subgroup analysis and multivariate regression analysis will be done.
* Adverse effects - No adverse effect is expected to occur out of the study protocol.
* Stopping rule - Not Valid

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing major HPB cancer surgeries at ILBS from 2010 till 30th June 2024.

Exclusion Criteria:

1. Presence of diuretic (Thiazide, Frusemide), pain killer (Indomethacin, Ketorolac) induced preoperative hyponatremia.
2. Patients with peri-operative diarrhea and vomiting due to infective cause leading to hyponatremia.
3. Patients who did not have a preoperative serum sodium level recorded within 72 hours prior to surgery.
4. Minor HPB cases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients undergoing major HPB surgery from 2010 till 30th June 2024.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Post operative major morbidities and early mortality (<90 day). | Post operative day 90
  Post operative major morbidities and early mortality (<90 day) in major HPB surgeries done for cancer. in patients with and without peri-operative hyponatremia. (<135mmoL/L).

SECONDARY OUTCOMES:
Post operative Systemic complications. | Post operative day 90
  Post operative Systemic complications in patients with and without peri-operative hyponatremia.
Overall Survival | Till 30th Sep 2024
  Overall Survival defined as POD1 till death/last follow up in patients with and without peri-operative hyponatremia.
Disease free survival | Till 30th Sep 2024
  Disease free survival- Surgical resection till first detected recurrence of cancer or last follow-up without recurrence with and without peri-operative hyponatremia.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided